CLINICAL TRIAL: NCT03358719
Title: A Phase 1 Study of DEC205mAb-NY ESO 1 Fusion Protein (CDX-1401) Given With Adjuvant Poly-ICLC in Conjunction With 5-Aza-2'Deoxycytidine (Decitabine) and Nivolumab in Patients With MDS or Low Blast Count AML
Brief Title: DEC-205/NY-ESO-1 Fusion Protein CDX-1401, Poly ICLC, Decitabine, and Nivolumab in Treating Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 49217; NCI-2017-02012 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 49217 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2017-11-13; First posted 2017-12-02 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Blasts 30 Percent or Less of Bone Marrow Nucleated Cells; Chronic Myelomonocytic Leukemia; High Risk Myelodysplastic Syndrome; Myelodysplastic Syndrome; Refractory Anemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Anemia, Refractory | interventions — Decitabine; Injections; Nivolumab; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (CDX-1401, poly ICLC, decitabine, nivolumab) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 intracutaneously and poly ICLC SC on day -14, on day 15 of courses 1-4, and then on day 1 of every 4 courses thereafter. Patients also receive nivolumab IV over 30 minutes on days 1 and 15 and decitabine IV over 1 hour on days 1-5. Courses with nivolumab and decitabine repeat every 4 weeks in the absence of disease progression or unaccepted toxicity.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Poly ICLC

INTERVENTIONS:
Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401 — Given intracutaneously
  Other Names: CDX-1401
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Drug: Poly ICLC — Given SC
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid

SUMMARY:
This phase I trial studies the side effects of DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, decitabine, and nivolumab in treating patients with myelodysplastic syndrome or acute myeloid leukemia. DEC-205/NY-ESO-1 fusion protein CDX-1401 is a vaccine that may help the immune system specifically target and kill cancer cells. Poly ICLC may help stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as nivolumab, may interfere with the ability of cancer cells to grow and spread. Giving DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, decitabine, and nivolumab may work better in treating patients with myelodysplastic syndrome or acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of NY-ESO-1 vaccination (Anti-DEC-205-NY-ESO-1 fusion protein + poly-ICLC) given in combination with decitabine 20 mg/m^2 intravenously and nivolumab 3 mg/kg in patients with myelodysplastic syndrome (MDS) or low blast count acute myeloid leukemia (AML).

SECONDRY OBJECTIVES:

I. Assess immune and molecular epigenetic responses following combination therapy with nivolumab, decitabine and NY-ESO-1 fusion protein CDX-1401 (NY-ESO-1) vaccination.

TERTIARY OBJECTIVES:

I. To record the response rate (complete response, partial response and hematological improvement) in MDS or low blast count AML patients treated with the combination in order to provide descriptive characteristics.

II. To record the overall survival (OS), progression free survival (PFS) and time to AML transformation (TTT) (for patients with MDS at diagnosis) enrolled on the study.

OUTLINE:

Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 intracutaneously and poly ICLC subcutaneously (SC) on day -14, on day 15 of courses 1-4, and then on day 1 of every 4 courses thereafter. Patients also receive nivolumab intravenously (IV) over 30 minutes on days 1 and 15 and decitabine IV over 1 hour on days 1-5. Courses with nivolumab and decitabine repeat every 4 weeks in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up at 30, 60, 90, and 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of:

  * International Prognostic Scoring System (IPSS) intermediate-1, intermediate-2 or high-risk MDS including chronic myelomonocytic leukemia (CMML) OR
  * Low blast count AML with =< 30% blasts previously classified as refractory anemia with excess blasts in transformation
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Hepatic:
* Total bilirubin =< 3 X upper limit of normal (ULN) (except subjects with Gilbert syndrome, who can have total bilirubin up to 3.5 X ULN)
* Aspartate aminotransferase (aspartate transaminase [AST]/serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (alanine transaminase [ALT]/serum glutamate pyruvate transaminase [SGPT]) =< 3 X ULN
* Serum creatinine =< 2.5 X ULN
* Troponin-I =< ULN
* Creatine kinase (CK)-MB =< ULN
* Left ventricular ejection fraction (LVEF) >= ULN (institutional limit)
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* No prior exposure to Nivolumab
* No prior investigational therapy within 2 weeks prior to study enrollment

Exclusion Criteria:

* We will exclude patients who are eligible for an allogeneic bone marrow transplant at the time of study enrollment; if an enrolled patient subsequently becomes eligible for transplant, they will not be prevented from proceeding to the appropriate clinical treatment indicated
* Subjects with life-threatening illnesses other than MDS, uncontrolled medical conditions or organ system dysfunction which, in the investigator?s opinion, could compromise the subject?s safety, or put the study outcomes at risk
* AML associated with inv(16); t(16;16); t(8;21) or t(15;17)
* Previously untreated MDS with isolated del5q (for which lenalidomide is approved as approved therapy) and chronic myelomonocytic leukemia (CMML) with rearrangements of the PDGF receptor (for which imatinib is approved therapy) unless they have previously failed these approaches
* Subjects with symptomatic central nervous system (CNS) disease which is not adequately controlled
* Subjects who have received prior radiation therapy for extramedullary disease within 2 weeks of first dose
* Has known immunosuppressive disease (e.g. human immunodeficiency virus [HIV], acquired immunodeficiency syndrome [AIDS] or other immune depressing disease); testing is not required, only to be done for a possible diagnosis which is not confirmed
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; in addition, subjects will be excluded for any of the following:

  * Myocardial infarction or arterial or venous thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) class III or IV disease
  * Active congestive heart failure (New York Heart Association functional classification III or IV)
  * Documented history of cardiomyopathy with EF < 30%
  * Uncontrolled hypertension (systolic blood pressure [SBP] > 160/diastolic blood pressure [DBP] > 100 despite medical intervention)
  * History of myocarditis of any etiology
* Subjects who have hypersensitivity to decitabine, CDX-1401, poly-ICLC or nivolumab
* History of auto-immune disease (e.g., thyroiditis, lupus), except vitiligo
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Regular use of immunosuppressant drugs such as steroids (> 20 mg prednisone equivalents), azathioprine, tacrolimus, cyclosporine, etc>. Use is not permitted within 4 weeks before recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 180 days
  Will evaluate the proportion of n=12 evaluable patients in the expansion cohort experiencing a dose-limiting toxicity. Toxicity rates will be described using upper 1-sided 95% Jeffreys binomial confidence intervals.

SECONDARY OUTCOMES:
Immune cell profile | Up to 180 days
  Descriptive statistics will be used to evaluate the Immune cell profile in the peripheral blood and bone marrow following combination therapy using mass cytometry.
Peripheral blood and bone marrow cells responses | Up to 180 days
  Will determine the impact of combination treatment on peripheral blood and bone marrow cells from patients treated in this manner on NY-ESO-1 target gene expression, NY-ESO-1 protein expression, NY-ESO-1 promoter methylation, and global deoxyribonucleic acid (DNA) methylation. The statistical significance of the change in marker values resulting from treatment will be assessed using the (paired sample) Wilcoxon Signed Rank test.

OTHER OUTCOMES:
Complete Response rate | Up to 180 days
  Will be assessed by complete response (CR), using results of blood counts on day 1 of each cycle.
Partial Response Rate | Up to 180 days
  Will be assessed by partial response (PR) using results of blood counts on day 1 of each cycle.
Hematologic Improvement | Up to 180 days
  Will be assessed by Hematologic Improvement using results of blood counts on day 1 of each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Griffiths, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Griffiths EA, Srivastava P, Gomez EC, Matsuzaki J, Odunsi K, Dillon LW, Mukherjee D, Hourigan CS, Peng J, Bandyopadhyay S, Tan K, Attwood KM, Kuechle JB, Singh PK, Wang J, Nemeth MJ. Checkpoint immunotherapy is associated with preferential activation of tumor antigen-specific CD4+ T cells in MDS. Blood Neoplasia. 2025 Apr 25;2(3):100106. doi: 10.1016/j.bneo.2025.100106. eCollection 2025 Aug. PMID 40809194